Study protocol: The Effect of Blood Pressure on Cerebral Blood Flow During

**Propofol Anesthesia** 

Brief Title: The Effect of Blood Pressure on Cerebral Blood Flow During Propofol Anesthesia

Official Title: The Effect of Blood Pressure on Cerebral Blood Flow During Propofol Anesthesia

Acronym: CA

Clinical trials ID: NCT03309917

Date: December 22 2017

**Unique Protocol ID:** H-17021598-61256

## **Ethics**

The study protocol (H-17021598-61256) was approved by the Regional Ethical Committee of the Copenhagen Region (De Videnskabsetiske Komiteer Region Hovedstaden, 004538666395, Email: <a href="https://www.wek.argeionh.dk">wek.argeionh.dk</a>, Adress: Kongens Vænge 2, DK-3400 Hillerød, Denmark

The study is monitored by the Danish Dataprotection Agency.

Study is planned to be conducted from December 2017-April 2018

FDA Regulated: No

FDA Regulated Intervention: No

Sponsor: Rigshospitalet, Denmark

Principal investigator: Niels Damkjær Olesen, MD

Sub-Investigator: Niels H. Secher, M.D., D.M.Sc., Prof.

# **Contacts/Locations**

## **Central Contact:**

Niels D. Olesen, MD

Telephone: 0045 35452674

Email: nielsdolesen@gmail.com

# **Central Contact Backup:**

Niels H. Secher, M.D., D.M.Sc., Prof..

Telephone: 0045 35452242

Email: niels.secher@regionh.dk

**Study Officials:** 

Niels D. Olesen, MD

Study Principal Investigator

Department of Anesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark

**Locations:** 

Department of Anesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark

Facility contact: Niels D. Olesen, M.D. Tel.: 0045 35452674 e-mail: nielsdolesen@gmail.com

**Short Description** 

General anesthesia often reduces blood pressure whereby blood flow to the brain and other vital organs may become insufficient. Thus, medicine is often administered to maintain blood pressure but it is unclear at what level blood pressure should be aimed at during anesthesia.

Thirty patients undergoing major abdominal surgery will be included. The study will start one hour after the start of surgery and lasts for approximately half an hour. The purpose of the study is to evaluate whether blood flow to the brain can be increased by maintaining blood pressure at a higher level than that used in clinical practice. In the study, MAP is adjusted to a high, moderate, and low level for a short time. The low level of blood pressure used in the study, corresponds to the level aimed at in clinical practice. The drug noradrenaline will be used to control blood pressure. Blood flow to the brain will be evaluated on the neck using ultrasound.

**Background** 

Propofol anesthesia reduces cerebral blood flow (CBF) and mean arterial pressure (MAP) but it is unclear whether the decrease in CBF is accentuated by hypotension. Cerebral autoregulation is

generally considered to maintain CBF when MAP is between 60-150 mmHg. Hence, vasoactive medication is administered if MAP decreases to below approximately 60 mmHg.

It is controversial whether there is a plateau for cerebral autoregulation. Thus, middle cerebral artery blood velocity (MCA Vmean), as an index of CBF, is associated to MAP during pharmacological changes in MAP between approximately 40-125 mmHg. Similarly, CBF is affected by pharmacological changes in MAP between 40-80 mmHg during hypothermic cardiopulmonary bypass surgery in propofol anesthesia. Arterial hypertension may increase the lower limit of cerebral autoregulation which can be mitigated by antihypertensive treatment.

Cognitive dysfunction and delirium are common following major surgery, particularly in the elderly, and may be related to hypotension and cerebral hypoperfusion. Further, hypotensive anesthesia is associated with an increase in markers of neuronal damage, but studies have been too small to detect any difference in incidence of cognitive dysfunction following hypotensive as compared to normotensive anesthesia.

In young healthy adults, propofol anesthesia causes limited reduction in blood pressure and decreases CBF by approximately 50% by a reduction in neuronal activity. An increase in MAP from approximately 80 to 100 mmHg during propofol anesthesia does not affect CBF but it is unknown whether CBF can be increased by an increase in MAP from approximately 60 to 80 mmHg. Propofol appears to maintain cerebral autoregulation but it is unknown whether the lower level of cerebral autoregulation is affected. The internal carotid artery supplies most of CBF and dilates during moderate hypotension with maintained blood flow which indicates that the vessel contributes to cerebral autoregulation. Further, central blood volume and cardiac output may be important factors for maintaining CBF.

The study will include thirty patients planned for major abdominal surgery in propofolremifentanil anesthesia combined with epidural analgesia. Internal carotid artery blood flow will be evaluated on the neck using duplex ultrasound. The study will be conducted one hour after the start of surgery and lasts for approximately half an hour. In the study, MAP is set pharmacologically at 80-85, 70-75 and 60-65 mmHg for a short time in random order. The level of 60-65 mmHg corresponds to the level at which MAP is maintained in clinical practice. Control of MAP is by intravenous infusion of noradrenaline, an  $\alpha$  - and  $\beta$  -adrenergic agonist.

# **Objective**

The purpose of the study is to evaluate whether internal carotid artery blood flow is increased by maintaining MAP at a higher level than that used in clinical practice during propofol anesthesia. Further, we evaluate whether a lower limit of cerebral autoregulation can be detected by comparing the slopes of linear regression of internal carotid artery blood flow and MAP at the evaluations when MAP is 60-65 and 70-75 mmHg and when MAP is 70-75 and 80-85 mmHg.

# **Hypotheses**

- Internal carotid artery blood flow is higher when MAP is 80-85 mmHg as compared to a MAP of 60-65 mmHg.
- Internal carotid artery blood flow is higher when MAP is 70-75 mmHg as compared to a MAP of 60-65 mmHg.
- Internal carotid artery blood flow is higher when MAP is 80-85 mmHg as compared to a MAP of 70-75 mmHg.
- The slope of linear regression between changes in MAP and internal carotid artery blood flow is higher for the evaluations at a MAP of 70-75 and 60-65 mmHg than for the evaluations at a MAP of 80-85 and 70-75 mmHg.

## **Methods**

The study is a single-center, prospective cohort study of thirty consecutive patients planned for major abdominal surgery in propofol anesthesia. In case surgery is cancelled, or if gas anesthesia is used the patient will be excluded and excluded patients will be replaced. The number of dropouts is expected to be between zero to five patients. Patients will be recruited the day before surgery, at which time the internal carotid artery will be evaluated using ultrasound. In case the vessel cannot be visualized, e.g. due to high localization of the carotid bifurcation the patient will not be able to participate in the study.

Anesthesia and surgery are according to clinical practice. Anesthesia is induced by propofol and maintained by propofol and remifentanil. A thoracic epidural catheter is placed at Th8/9 or Th9/10 and epidural anesthesia is initiated before surgery by bupivacaine infusion 0.5%, 5 ml/hr. and bolus 15 mg bupivacaine that is repeated hourly. Stroke volume is optimized after induction of anesthesia by repeated administration of 250 ml 5% human albumin until the increase in stroke volume is less than 10%, and volume optimization is repeated in case of persistent decrease in stroke volume by more than 10%. Noradrenaline infusion (0.6  $\mu$  g/kg\*ml) is started after induction of anesthesia to maintain MAP > 60 mmHg and to avoid volume optimization when the circulation is dilated.

Development of a so-called mesenteric traction syndrome can affect MAP in the first hour of major abdominal surgery. Thus, the study is conducted from 60 min after incision and lasts for approximately half an hour. Anesthesia reduces MAP, but the reduction varies between patients and is affected by administration of propofol, remifentanil, and epidural anesthesia, fluid status, and surgical stimulation etc. The start of the study is postponed until any larger bleeding, transfusion or volume optimization is treated or finished. Before the start of the study, the infusion speed of propofol and remifentanil must have been constant for at least 10 min, and at least 15 min must have elapsed since the last bolus dose bupivacaine, as any changes in anesthesia may affect both

cerebral and central hemodynamics. In case the infusion of propofol or remifentanil is changed or bolus bupivacaine is administered during the study, the experiment is halted, and the study is restarted when the anesthesia has been stable for 10 min. The experiment can only be restarted once and only data from the last trial with the highest number of evaluations are used.

In the experiment MAP is temporally set to 80-85, 70-75, and 60-65 mmHg by adjusting the infusion of noradrenaline. The order of evaluations is randomized by drawing an envelope just before the start of the experiment. Noradrenaline is short lasting and have no direct effect on CBF. The experiment lasts approximately 30 min until evaluations have been conducted at the three levels of MAP. If MAP does not drop to 60-65 mmHg by halting the infusion of noradrenaline this evaluation is not conducted but we expect that this will be the case in only few patients. In clinical practice noradrenaline is used to maintain MAP > 60 mmHg. The study is not an investigation of medicinal products as noradrenaline is used as a tool to control MAP.

Administration of noradrenaline is by a central venous or large peripheral catheter, using an electronic infusion pump, and infusion speed is adjusted slowly until the level of MAP is reached. Noradrenaline is effective within 1-2 min after administration and the effect lasts only for a few minutes. When MAP has been stable at the desired level for at least 3 min, measurements are conducted during the following 2 min. When the study is finished, control of MAP will be according to clinical practice. We consider that there is no increased risk by a short term increase in MAP to 80-85 mmHg.

#### Measurements

Arterial and central venous pressure are determined invasively while stroke volume, cardiac output, and total peripheral resistance are evaluated by modified pulse-contour analysis of the arterial pressure curve (Nexfin, BMEYE, Holland). Cerebral and biceps muscle oxygenation are evaluated

using near-infrared spectroscopy (INVOS 5100C, Somanetics, Troy, MI, USA). Depth of anesthesia is assessed by Bispectral Index (BIS Complete Monitoring Systems, Covidien, USA).

Internal carotid artery blood flow is evaluated unilaterally on the neck using duplex ultrasound (Logiq E, GE Medical System, Jiangsu, Kina). Evaluation is in the longitudinal section at least 1.5 cm distal to the carotid bifurcation with the head turned approximately  $30^{\circ}$  to the contralateral side. In order to limit the influence of ventilation, three recordings of approximately 15-20 s are conducted at each level of MAP and the mean is reported. A frequency of 8-12 MHz is used and gain is set as high as possible while vessel lumen is echo-free. Ultrasonic adjustments are not changed during the study. Diameter is assessed using automatic software to track the vessel wall (Brachial Analyser for Research v. 6, Medical Imaging Applications LLC, Coralville, IA, USA). The angle-corrected time maximum flow velocity (TAVMAX) is evaluated using pulsed-wave Doppler at an angle of insonation  $\leq 60^{\circ}$ . The TAVMAX corresponds to twice the mean blood velocity and blood flow is:  $0.125*60*TAVMAX*\pi*$ diameter^2. Arterial and central venous blood is sampled for blood gas analysis. Internal carotid artery blood flow is corrected for changes in PaCO<sub>2</sub> using a factor of 18%/kPa and for the  $S_cO_2$  a correction factor of 4.3%/kPa is used (unpublished results from the study "Cerebral Blood Flow During Propofol Anaesthesia" NCT02951273).

## **Statistics**

Trial size: The minimal clinically important difference in internal carotid artery blood flow between evaluations at MAP 60-65 and 80-85 mmHg is considered to be 10% as evaluations using near-infrared spectroscopy indicate that intraoperative cerebral deoxygenation of > 10% associates to postoperative cognitive dysfunction.

A power calculation indicated that at least 18 patients were required to detect a difference in internal carotid artery blood flow of 10% corresponding to 19 ml/min assuming a standard deviation for the change of 27 ml/min (unpublished results from the study "Cerebral Blood Flow During Propofol Anaesthesia" NCT02951273) to obtain a 5% significance level and a power of 80%. We plan to include 30 patients.

# **Inclusion Criteria**

- Patient planned for Whipple's surgery or total pancreatic resection
- Age > 18 years

# **Exclusion Criteria**

- No informed consent
- Alcohol intake  $\geq 420 \text{ g}$  / week
- Beard on the neck
- Visualization of the internal carotid artery not possible, e.g. due to high
- placement of the bifurcation
- Stenosis that obstructs  $\geq 16\%$  of the internal carotid artery
- Cardiac disease, including congestive heart failure (NYHA II-IV),
- myocardial infarction, valvular heart disease or atrial fibrillation
- Neurologic disease considered to affect cerebral blood flow, including
- dementia, epilepsy, and apoplexy

 Intake of moclobemide, isocarboxazid or tricyclic antidepressantsNeurologic disease considered

# **Primary Outcome Measure:**

 Change in internal carotid artery blood flow when mean arterial pressure (MAP) is set to 80-85 and 60-65 mmHg

# **Secondary Outcome Measures:**

- 2. Change in internal carotid artery blood flow when MAP is set to 70-75 and 60-65 mmHg
- 3. Change in internal carotid artery blood flow when MAP is set to 80-85 and 70-75 mmHg
- 4. Comparison of the slope of linear regression of MAP and internal carotid artery blood flow for the evaluations when MAP is set to 80-85 and 70-75 mmHg and that of the evaluations when MAP is set to 70-75 and 60-65 mmHg

## References

Choi WS, Samman N. Risks and benefits of deliberate hypotension in anaesthesia: a systematic review. Int J Oral Maxillofac Surg. 2008;37:687-703.

Ederberg S, Westerlind A, Houltz E, Svensson SE, Elam M, Ricksten SE. The effects of propofol on cerebral blood flow velocity and cerebral oxygen extraction during cardiopulmonary bypass. Anesth Analg. 1998;86:1201-6.

Evans DH. On the measurement of the mean velocity of blood flow over the cardiac cycle using Doppler ultrasound. Ultrasound Med Biol. 1985;11:735-41.

Greenfield JC, Jr., Tindall GT. Effect of norepinephrine, epinephrine, and angiotensin on blood flow in the internal carotid artery of man. J Clin Invest. 1968;47:1672-84.

Jiang X, Chen D, Lou Y, Li Z. Risk factors for postoperative delirium after spine surgery in middleand old-aged patients. Aging Clin Exp Res. 2016. Jørgensen LG, Perko M, Perko G, Secher NH. Middle cerebral artery velocity during head-up tilt induced hypovolaemic shock in humans. Clin Physiol. 1993;13:323-36.

Kaisti KK, Langsjo JW, Aalto S, Oikonen V, Sipila H, Teras M, et al. Effects of sevoflurane, propofol, and adjunct nitrous oxide on regional cerebral blood flow, oxygen consumption, and blood volume in humans. Anesthesiology. 2003;99:603-13.

Kaisti KK, Metsahonkala L, Teras M, Oikonen V, Aalto S, Jaaskelainen S, et al. Effects of surgical levels of propofol and sevoflurane anesthesia on cerebral blood flow in healthy subjects studied with positron emission tomography. Anesthesiology. 2002;96:1358-70.

Kety SS, King BD, Horvath SM, Jeffers WS, Hafkenschiel JH. The effects of an acute reduction in blood pressure by means of differential spinal sympathetic block on the cerebral circulation of hypertensive patients. J Clin Invest. 1950;29:402-7.

Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, et al. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014;35:2383-431.

Lassen NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959;39:183-238.

Li S, Hoskins PR, Anderson T, McDicken WN. Measurement of mean velocity during pulsatile flow using time-averaged maximum frequency of Doppler ultrasound waveforms. Ultrasound Med Biol. 1993;19:105-13.

Lin R, Zhang F, Xue Q, Yu B. Accuracy of regional cerebral oxygen saturation in predicting postoperative cognitive dysfunction after total hip arthroplasty: regional cerebral oxygen saturation predicts POCD. J Arthroplasty. 2013;28:494-7.

Lin S, McKenna SJ, Yao CF, Chen YR, Chen C. Effects of Hypotensive Anesthesia on Reducing Intraoperative Blood Loss, Duration of Operation, and Quality of Surgical Field During Orthognathic Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2017;75:73-86.

Liu J, Zhu YS, Hill C, Armstrong K, Tarumi T, Hodics T, et al. Cerebral autoregulation of blood velocity and volumetric flow during steady-state changes in arterial pressure. Hypertension. 2013;62:973-9.

Lucas SJ, Tzeng YC, Galvin SD, Thomas KN, Ogoh S, Ainslie PN. Influence of changes in blood pressure on cerebral perfusion and oxygenation. Hypertension. 2010;55:698-705.

Matta BF, Lam AM, Strebel S, Mayberg TS. Cerebral pressure autoregulation and carbon dioxide reactivity during propofol-induced EEG suppression. Br J Anaesth. 1995;74:159-63.

Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015;123:1198-208.

Mille T, Tachimiri ME, Klersy C, Ticozzelli G, Bellinzona G, Blangetti I, et al. Near infrared spectroscopy monitoring during carotid endarterectomy: which threshold value is critical? Eur J Vasc Endovasc Surg. 2004;27:646-50.

Newman MF, Croughwell ND, Blumenthal JA, White WD, Lewis JB, Smith LR, et al. Effect of aging on cerebral autoregulation during cardiopulmonary bypass. Association with postoperative cognitive dysfunction. Circulation. 1994;90:II243-9.

Newman S, Stygall J, Hirani S, Shaefi S, Maze M. Postoperative cognitive dysfunction after noncardiac surgery: a systematic review. Anesthesiology. 2007;106:572-90.

Olesen J. The effect of intracarotid epinephrine, norepinephrine, and angiotensin on the regional cerebral blood flow in man. Neurology. 1972;22:978-87.

Olesen J. Beta-adrenergic effects on cerebral circulation. Cephalalgia : an international journal of headache. 1986;6 Suppl 5:41-6.

Olesen J, Paulson OB, Lassen NA. Regional cerebral blood flow in man determined by the initial slope of the clearance of intra-arterially injected 133Xe. Stroke. 1971;2:519-40.

Olesen ND, Sorensen H, Ambrus R, Svendsen LB, Lund A, Secher NH. A mesenteric traction syndrome affects near-infrared spectroscopy evaluated cerebral oxygenation because skin blood flow increases. J Clin Monit Comput. 2017:doi: 10.1007/s10877-017-0014-2.

Panerai RB. Assessment of cerebral pressure autoregulation in humans--a review of measurement methods. Physiol Meas. 1998;19:305-38.

Patti R, Saitta M, Cusumano G, Termine G, Di Vita G. Risk factors for postoperative delirium after colorectal surgery for carcinoma. Eur J Oncol Nurs. 2011;15:519-23.

Rollason WN, Robertson GS, Cordiner CM, Hall DJ. A comparison of mental function in relation to hypotensive and normotensive anaesthesia in the elderly. Br J Anaesth. 1971;43:561-6.

Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, et al. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011;40:200-7.

Sieskiewicz A, Groblewska M, Lyson T, Piszczatowski B, Turek G, Rutkowski R, et al. Neurobiochemical markers of brain ischemia in patients subjected to endoscopic skull base surgery under controlled hypotension. J Neurosurg Sci. 2016;60:313-9.

Song XX, Yu BW. Anesthetic effects of propofol in the healthy human brain: functional imaging evidence. J Anesth. 2015;29:279-88.

Strandgaard S. Autoregulation of cerebral blood flow in hypertensive patients. The modifying influence of prolonged antihypertensive treatment on the tolerance to acute, drug-induced hypotension. Circulation. 1976;53:720-7.

Strebel S, Lam AM, Matta B, Mayberg TS, Aaslid R, Newell DW. Dynamic and static cerebral autoregulation during isoflurane, desflurane, and propofol anesthesia. Anesthesiology. 1995;83:66-76.

Strebel SP, Kindler C, Bissonnette B, Tschaler G, Deanovic D. The impact of systemic vasoconstrictors on the cerebral circulation of anesthetized patients. Anesthesiology. 1998;89:67-72.

Thomas KN, Lewis NC, Hill BG, Ainslie PN. Technical recommendations for the use of carotid duplex ultrasound for the assessment of extracranial blood flow. Am J Physiol Regul Integr Comp Physiol. 2015;309:R707-20.

Torella F, McCollum CN. Regional haemoglobin oxygen saturation during surgical haemorrhage. Minerva Med. 2004;95:461-7.

Townes BD, Dikmen SS, Bledsoe SW, Hornbein TF, Martin DC, Janesheski JA. Neuropsychological changes in a young, healthy population after controlled hypotensive anesthesia. Anesth Analg. 1986;65:955-9.

Willie CK, Macleod DB, Shaw AD, Smith KJ, Tzeng YC, Eves ND, et al. Regional brain blood flow in man during acute changes in arterial blood gases. J Physiol. 2012;590:3261-75.